CLINICAL TRIAL: NCT00319761
Title: The Safety and Short-Term Efficacy of Calcitriol in the Treatment of Immunoglobulin A Nephropathy
Brief Title: Calcitriol in the Treatment of Immunoglobulin A (IgA) Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr. CC Szeto, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC-2006.120
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: IGA Nephropathy
Keywords: glomerulonephritis; proteinuria; chronic kidney diseases
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulonephritis; Proteinuria; Renal Insufficiency, Chronic | interventions — Calcitriol

INTERVENTIONS:
Drug: Calcitriol

SUMMARY:
Immunoglobulin A (IgA) nephropathy is the most common type of primary glomerulonephritis in the world. A wealth of literature suggests that vitamin D and its analogs have profound effects on immune system function and glomerular mesangial cell proliferation. Calcitriol, an active form of vitamin D, is commonly used for the treatment of secondary hyperparathyroidism in patients with advanced chronic kidney diseases. Therefore, the investigators plan to conduct a open-label single-arm study to evaluate the safety and efficacy of calcitriol in the treatment of IgA nephropathy. Ten patients with biopsy-proven IgA nephropathy and persistent proteinuria despite conventional therapy will be recruited. They will be treated with calcitriol for 12 weeks. Proteinuria, renal function, serum and urinary inflammatory markers will be monitored. This study will explore the potential anti-proteinuric and anti-inflammatory effects of calcitriol in the treatment of IgA nephropathy, which is a major cause of dialysis-dependent renal failure.

DETAILED DESCRIPTION:
This is a open-label and single arm study. We plan to recruit 10 patients with biopsy-proven IgA nephropathy will be recruited.

Treatment regimen and dosage adjustment

At week 0, all patients will receive calcitriol (oral capsule) at a fixed dose of 0.5 mcg twice weekly. If there is no adverse effect and corrected serum calcium remains < 2.55 mmol/l, the dose of calcitriol will be maintained for 12 weeks.

If corrected serum calcium is 2.55 to 2.62 mmol/l, the dose of calcitriol will be reduced to 0.25 mcg twice weekly. Serum calcium will be rechecked after 2 weeks (or more frequently if indicated). If corrected serum calcium remains < 2.55 mmol/l, the dose of calcitriol will be maintained for the rest of the study period. If corrected serum calcium remains > 2.62 mmol/l for two consecutive measurements despite reducing the dose of calcitriol, the study medication will be stopped and the subject will be discontinued from the study.

If corrected serum calcium is > 2.75 mmol/l at any time, hold calcitriol for one week and repeat laboratory test for calcium. If the subject's next serum calcium is < 2.62 mmol/l, calcitriol may be restarted at 0.25 mcg twice weekly. If the next serum calcium level is > 2.62 mmol/l, the subject will be discontinued from the study.

Concomitant therapy

Prior to enrollment, all of the patients will be stable while receiving ACE inhibitor or angiotensin receptor blocker. Anti-hypertensive therapy will be titrated throughout the study period to maintain the blood pressure below 130 / 80 mmHg.

Visit schedule

Follow up visits will take place according to the following schedule:

* week -4 (screening)
* weeks 0 (start calcitriol), 2, 4, 6, 8, 12 (stop calcitriol) and 16

During every visit, the following parameters will be measured: body weight, blood pressure, pulse, adverse effects of treatment, complete blood picture, differential white cell count, renal function test, liver enzymes, serum calcium, phosphate, and early morning urine collection for protein-to-creatinine ratio. Renal function is determined by the estimated glomerular filtration rate (GFR) according to a standardized formula [20]. Serum fasting glucose and lipid profile will be measured at 0 and 12 weeks.

In order to examine the anti-proliferative and anti-inflammatory action of calcitriol, serum level of C-reactive protein (CRP), interleukin-6 (IL-6) and transforming growth factor-beta (TGF), and urinary levels of TGF, hepatocyte growth factor (HGF), monocyte chemoattractant protein-1 (MCP-1) and thrombospondin-1 (TSP-1) will be measured at 0, 4, 12 and 16 weeks by ELISA. The above panel of cytokine is chosen because of their documented relevance in IgA nephropathy and progressive renal failure [16,19,21-27].

End points

Primary end point of the study is the change in the degree of proteinuria. Secondary end points include the change in renal function and other serum inflammatory markers.

Adverse events

Information about every adverse event will be collected and recorded. An adverse event is any undesirable symptom or medical condition occurring after starting the study medication, whether considered drug-related or not.

Patient withdrawal

The patient will be withdrawn from the study for:

* death
* doubling of baseline serum creatinine level
* pregnancy
* hypercalcemia (serum calcium > 2.62 mmol/L for two consecutive measurements)
* any other intolerable adverse events
* significant non-compliance with the protocol
* the desire of the patient to withdraw from the study All female patients will be advised on taking effective contraceptive measures during the study period.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* biopsy-confirmed IgA nephropathy
* proteinuria > 1 g/day (or proteinuria > 1 g/g-Cr) in 2 consecutive samples within 12 weeks despite ACE inhibitor or angiotensin receptor blocker treatment (ramipril 5 mg daily, lisinopril 10 mg daily, or valsartan 80 mg daily) for at least 3 months
* estimated glomerular filtration rate 15 to 60 ml/min/1.73m2
* corrected serum calcium level M 2.45 mmol/l
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* History of malignancy, including leukemia and lymphoma within the past 2 years
* Systemic infection requiring therapy at study entry
* Any other severe coexisting disease such as, but not limited to, chronic liver disease, myocardial infarction, cerebrovascular accident, malignant hypertension
* History of drug or alcohol abuse within past 2 years
* Participation in any previous trial on vitamin D analogue
* Patients receiving treatment of vitamin D and/or its analogue for other medical reasons within the past 3 months
* Patients receiving treatment of corticosteroid
* On other investigational drugs within last 30 days
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance
* Known history of sensitivity or allergy to vitamin D analogs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Primary end point of the study is the change in the degree of proteinuria.

SECONDARY OUTCOMES:
Secondary end points include the change in renal function and other serum inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk-Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Szeto CC, Chow KM, Kwan BC, Chung KY, Leung CB, Li PK. Oral calcitriol for the treatment of persistent proteinuria in immunoglobulin A nephropathy: an uncontrolled trial. Am J Kidney Dis. 2008 May;51(5):724-31. doi: 10.1053/j.ajkd.2007.12.038. Epub 2008 Apr 3. PMID 18436082